CLINICAL TRIAL: NCT01593982
Title: Effect of Repetitive Transcranial Magnetic Stimulation on Symptoms of Attention Deficit Hyperactivity Disorder and Cognitive Function In Cocaine Addicts
Brief Title: Repetitive Transcranial Magnetic Stimulation in Symptoms of Attention Deficit Hyperactivity Disorder and Cognitive Function In Cocaine Addicts
Acronym: rTMSinADHD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0181/08
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Cognition Disorders; Cocaine Dependence; ADHD
Keywords: Repetitive Transcranial Magnetic Stimulation; Cocaine Dependence; Cocaine Addicts; Attention Deficit Hyperactivity Disorder; Cognitive Function
MeSH Terms: conditions — Cognition Disorders; Cocaine-Related Disorders; Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham rTMS (Placebo Comparator): Drug-free patients, receiving 20 sessions (1 session daily) of Sham (placebo) rTMS delivered to the left dorsolateral prefrontal cortex.
  Interventions: Other: repetitive Transcranial Magnetic Stimulation (rTMS)
- Active rTMS (Active Comparator): Drug-free patients, receiving 20 sessions (1 session daily) of Active rTMS delivered to the left dorsolateral prefrontal cortex.
  Interventions: Other: repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Other: repetitive Transcranial Magnetic Stimulation (rTMS) — 20 daily sessions: each with 25 trains of 10 seconds at 5Hz, with a 20 second inter-train interval, at an intensity of 120% of motor threshold.
  Site: Left Dorsolateral Prefrontal Cortex
  Other Names: TMS

SUMMARY:
Even in the absence of a preliminary diagnosis of Attention Deficit Hyperactivity Disorder, symptoms of attention deficit, hyperactivity and cognitive impairment are common in cocaine addicts.

Several factors indicate that repetitive transcranial magnetic stimulation might be a strategy to aid in the treatment of symptoms of attention deficit hyperactivity disorder and cognitive function in cocaine addicts.

However, up to current days there have been no studies evaluating the effects of Repetitive Transcranial Magnetic Stimulation (rTMS) on neurocognitive performance of individuals suffering from the ADHD.

DETAILED DESCRIPTION:
Transcranial Magnetic Stimulation is a noninvasive technique that can influence specific areas of the brain and has very few side effects.

The treatment with transcranial magnetic stimulation requires attendance to hospital daily sessions for 4 consecutive weeks. Each session lasts up to 30 minutes.

Side effects include scalp discomfort and mild headache. No anesthesia is required.

Stimulation aims the dorsolateral prefrontal cortex, a region previously studied to treat depression symptoms with positive results.

The present technique has never been employed in previous studies, but risks are insignificant.

ELIGIBILITY:
Inclusion Criteria:

* Cocaine Dependence Syndrome (alone or in combination with alcohol and/or nicotine dependence with symptoms of ADHD, according to the criteria of the DSM-IV-R (APA, 2000), as well as through a structured clinical interview (SCID-1/P v 2.0)
* Minimum age of 18
* Maximum age of 40
* 20 days or less abstinence.
* any psychopharmacological treatment other than clonazepam (4 mg/day)

Exclusion Criteria:

* Metallic Cerebral Implant
* Pacemakers
* History of Severe Brain trauma or injury
* Organic Brain Disease
* Previous neurosurgery
* History of seizures
* Epilepsy
* Severe Somatic Disease
* History of other actual or past psychiatric diagnostics
* Clinically significant changes in laboratory test
* Any psychiatric or neurological disorder other than Cocaine Dependence with symptoms of ADHD
* Psychotic depression
* Suicidal propensities

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-08 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Wender Utah Rating Scale (WURS) - Diagnostic Criteries ADHD (DSM IV) | 4 weeks
  Scales to assess attention deficit hyperactivity disorder symptoms will be applied at pre-treatment (T0) and post treatment - week 4 (T1).
  Reduction on the scores of WURS and synptoms of ADHD diagnostic (as on the scores of Barrat Impulsiviness Scale - BIS 11 and Minnesota Cocaine Craving Scale - MCCS; and improves Hamilton Depressive Rating Scale - HDRS 17 and Hamilton Anxiety Rating Scale - HARS 14).

SECONDARY OUTCOMES:
Battery of Neuropsychological Tests | 4 weeks
  Cognitive performance battery will be applied at pre-treatment (T0) and post treatment - week 4 (T1).
  Performance of neuropsychological tests - Trail Making Test; Wisconsin Card Sorting Test; Controlled Oral Word Association Test; Victoria Stroop Test; Rey Auditory Verbal Learning Test; WAIS-III (adapted for use in Brazil) subtests Cubes, Vocabulary, Digit Span; Wechsler Logical Memory and Iowa Gambling Task (IGT).

CONTACTS AND LOCATIONS:
Overall Officials: Debora Arnaut, PSYD, Principal Investigator — Laboratory of Brain Stimulation - Institute of Psychiatry, General Hospital, University of Sao Paulo Medical School
Locations (1):
- Department and Institute of Psychiatry, General Hospital, University of Sao Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] van Emmerik-van Oortmerssen K, van de Glind G, van den Brink W, Smit F, Crunelle CL, Swets M, Schoevers RA. Prevalence of attention-deficit hyperactivity disorder in substance use disorder patients: a meta-analysis and meta-regression analysis. Drug Alcohol Depend. 2012 Apr 1;122(1-2):11-9. doi: 10.1016/j.drugalcdep.2011.12.007. Epub 2011 Dec 30. PMID 22209385
- [Background] Gudjonsson GH, Sigurdsson JF, Sigfusdottir ID, Young S. An epidemiological study of ADHD symptoms among young persons and the relationship with cigarette smoking, alcohol consumption and illicit drug use. J Child Psychol Psychiatry. 2012 Mar;53(3):304-12. doi: 10.1111/j.1469-7610.2011.02489.x. Epub 2011 Nov 8. PMID 22066497
- [Background] Bloch Y, Harel EV, Aviram S, Govezensky J, Ratzoni G, Levkovitz Y. Positive effects of repetitive transcranial magnetic stimulation on attention in ADHD Subjects: a randomized controlled pilot study. World J Biol Psychiatry. 2010 Aug;11(5):755-8. doi: 10.3109/15622975.2010.484466. PMID 20521875
- [Background] Barr MS, Farzan F, Wing VC, George TP, Fitzgerald PB, Daskalakis ZJ. Repetitive transcranial magnetic stimulation and drug addiction. Int Rev Psychiatry. 2011 Oct;23(5):454-66. doi: 10.3109/09540261.2011.618827. PMID 22200135